CLINICAL TRIAL: NCT07152600
Title: An Embedded Adaptive Randomized Controlled Trial of Corticosteroid Therapy for Severe Adenovirus Community-Acquired Pneumonia in Adults
Brief Title: Adaptive RCT of Corticosteroids for Severe Adenovirus Pneumonia in Adults
Acronym: CAPSTONE-AD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qingyuan Zhan (Other)
Responsible Party: Sponsor-Investigator, Qingyuan Zhan, Director, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-I2M-C&T-B-090A
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Adenovirus Infections, Human
Keywords: Adenovirus; community-acquired pneumonia; adaptive randomised controled trial; corticosteroids
MeSH Terms: conditions — Adenovirus Infections, Human; Adenoviridae Infections; Community-Acquired Pneumonia | interventions — Sodium Chloride; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Placebo Comparator): Control group
  Interventions: Drug: Saline (0.9%, sterile, for infusion)
- Low dose steroids (Experimental): treated with low dose corticosteroids
  Interventions: Drug: low dose Methylprednisolone
- Moderate dose steroids (Experimental): treated with moderate dose corticosteroids
  Interventions: Drug: Moderate dose Methylprednisolone

INTERVENTIONS:
Drug: Saline (0.9%, sterile, for infusion) — Sailine as control
  Arms: Standard of Care
Drug: low dose Methylprednisolone — Methylprednisolone 0.5mg/kg ivgtt qd
  Arms: Low dose steroids
Drug: Moderate dose Methylprednisolone — Methylprednisolone 1.0mg/kg ivgtt qd
  Arms: Moderate dose steroids

SUMMARY:
Severe community-acquired pneumonia caused by adenovirus (hereafter referred to as severe adenovirus pneumonia) is one of the common forms of severe community-acquired pneumonia in immunocompetent adults. It predominantly affects young individuals, progresses rapidly, and is associated with a high incidence of respiratory failure and multiple organ dysfunction. At present, there is no effective antiviral therapy available in China, and the reported mortality rate ranges from 41.5% to 80%. How to effectively reduce the mortality of severe adenovirus pneumonia, on the basis of conventional supportive care, is crucial for improving the prognosis of critically ill patients and alleviating the burden on families and society. We are currently conducting an adaptive, randomized, open-label controlled trial aimed at reducing mortality in severe adenovirus pneumonia. The primary objective of this study is to evaluate the efficacy and safety of adjunctive corticosteroid therapy at different dosages, in addition to early standard supportive treatment, in lowering mortality among patients with severe adenovirus pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Admission to the Intensive Care Unit (ICU).
* Meeting the diagnostic criteria for community-acquired pneumonia (CAP).
* Meeting at least one of the major diagnostic criteria for severe pneumonia:

  (i) Requirement for endotracheal intubation and mechanical ventilation;

(ii) Septic shock requiring vasopressor therapy after adequate fluid resuscitation.

-Or simultaneously fulfilling three of the minor criteria:

(i) Respiratory rate ≥ 30 breaths/min;

(ii) PaO₂/FiO₂ ≤ 250 mmHg;

(iii) Multilobar infiltrates;

(iv) Altered mental status and/or disorientation;

(v) Blood urea nitrogen ≥ 20 mg/dL (7.12 mmol/L);

(vi) Leukopenia (white blood cell count < 4 × 10⁹/L);

(vii) Thrombocytopenia (platelet count < 100 × 10⁹/L);

(viii) Hypothermia (core temperature < 36 °C);

(ix) Hypotension (systolic blood pressure < 90 mmHg) requiring aggressive fluid resuscitation.

* Confirmed adenovirus etiology: at least one positive nucleic acid test (PCR) or next-generation sequencing (NGS) result for adenovirus in respiratory specimens (respiratory secretions, throat swabs, or bronchoalveolar lavage fluid).
* Severe community-acquired pneumonia (SCAP) patients admitted to the emergency department/ward/ICU due to respiratory failure within < 72 hours.
* Signed informed consent.

Exclusion Criteria:

* Patients receiving vasopressor therapy for septic shock at the time of enrollment.
* Terminally ill patients (expected survival <30 days, e.g., advanced malignancy).
* Clinical history suggesting overt aspiration.
* Documented active gastrointestinal bleeding.
* Presence of cystic fibrosis, obstructive pneumonia, active influenza, pulmonary tuberculosis, or fungal infection.
* Active viral hepatitis or active herpesvirus infection.
* Bone marrow suppression or HIV infection.
* Refusal of mechanical ventilation and endotracheal intubation.
* Uncontrolled hyperglycemia (diabetic ketoacidosis with blood ketones >3 mmol/L, or hyperosmolar hyperglycemic state with blood glucose >33.3 mmol/L and elevated osmolality).
* Known allergy to corticosteroids.
* Patients requiring anti-inflammatory corticosteroids or replacement hydrocortisone for any reason, or those already receiving prednisone >15 mg/day (or equivalent dose of another corticosteroid).
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day all cause mortality | 28 days from inclusion

IPD SHARING:
Plan to Share IPD: Undecided